CLINICAL TRIAL: NCT01079000
Title: Emergency Department (ED)-Directed Interventions to Improve Outcomes After Asthma Exacerbations
Brief Title: Emergency Department (ED)-Directed Interventions to Improve Asthma Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR operating grant # 201109; CIHR Grant (Other Grant/Funding Number: CIHR 201109 Operating Grant (MOP 119354))
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Acute Asthma
Keywords: asthma; exacerbation; emergency department; relapse
MeSH Terms: conditions — Asthma; Emergencies; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control - usual care (UC) (Active Comparator): Usual care after an ED visit for asthma will include the provision of discharge instructions/plan, and action plan, and verbal instructions for follow-up with their PCP, and a faxed copy of the ED chart to the patient's PCP.
  Interventions: Behavioral: Usual care
- Opinion leader (OL) guidance to patients' PCPs (Experimental): In addition to UC, OL guidance will be provided to the patients' PCP. A letter signed by an influential, respected, and local clinical leader (Respirologist) will encourage follow-up within two weeks and provide management suggestions.
  Interventions: Behavioral: Opinion Leader letter; Behavioral: Usual care
- Care manager education to patients (Experimental): In addition to UC and OL guidance provided to the patients' PCP, care manager self-management education will be provided to patients. A care manager will encourage patients' to pursue follow-up, provide management review and offer brief education via telephone within a week of being discharged.
  Interventions: Behavioral: Opinion Leader letter; Behavioral: Involvement of a care manager; Behavioral: Usual care

INTERVENTIONS:
Behavioral: Opinion Leader letter — The patients' PCP will be notified by fax about the ED visit and management. The Opinion Leader letter will contain a summary of the current asthma guidelines for ambulatory care (including: asthma education, long-term recommendations, smoking cessation, and action plan) signed by a local opinion leader. A review of the patient's management within a week of the ED visit will be recommended. The patient will also receive information regarding their acute exacerbation and will be told to review the current management of their disease with their PCP.
  Arms: Care manager education to patients; Opinion leader (OL) guidance to patients' PCPs
Behavioral: Involvement of a care manager — The involvement of a care manager will encourage patients' to pursue follow-up, provide management review and offer brief education via telephone within a week of being discharged
  Arms: Care manager education to patients
Behavioral: Usual care — Usual care provided to asthma patients when discharged from the ED

SUMMARY:
The purpose of this study is to determine if evidence-based guidance on follow-up care and self-management provided to PCPs and patients, respectively, reduces relapses within 90 days for acute asthma (primary outcome). Secondary outcomes will include follow-up visits with the primary care provider, patients' quality of life and cost-effectiveness indicators.

DETAILED DESCRIPTION:
This prospective, randomized, open label study will include asthmatics 17-55 years of age with no evidence of chronic obstructive pulmonary disease. Patients will be eligible if they visit one of four Emergency Departments (EDs) in Edmonton or Calgary and receive treatment for acute asthma resulting in discharge home. All patients should have a primary care provider (PCP: Family Physician, Internist or Nurse Practitioner) with whom to follow-up or one will be found for them. At discharge patients will be randomized into three groups: A: Usual care; PCPs will receive a faxed copy of the ED chart and patients will receive a discharge plan and a paper-based educational pamphlet (treatment in the ED and at discharge will be left to ED physicians' discretion); B: Usual care + personalized fax to the patients' PCP including a copy of the ED chart and a opinion-leader (OL) letter encouraging follow-up within two weeks and providing management suggestions; or C: Usual care + personalized fax to the patients' PCP including the OL letter as described above + involvement of a case manager who will encourage patients' to pursue follow-up, provide management review and offer brief education within the next week. Outcomes will be ascertained blinded to treatment allocation through telephone follow-up at 30 and 90 days. A sample of 366 patients (122 per group) is required based on the proportion with relapse at 90 days (40%) and a chi-square test of association and post-hoc tests (groups A vs. B, groups B vs. C). This sample will allow for the detection of an moderate effect size of at least 0.171, and a difference between groups A and B of 50% (i.e., 40% vs. 20%) and between groups B and C of 75% (i.e., 20% vs. 5%) using two-sided z-tests, 80% power, α=0.025. Intention to treat analyses will be conducted. Relapse rates by group and associated 95% confidence intervals (CI) will be calculated. Proportions among groups will be compared using chi-square tests and if statistically significant, separate proportion tests will compare pairs of groups adjusting for multiple testing. A multivariable logistic regression model will adjust effect estimates for potential baseline imbalances and site-specific differences in effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age 17-55 years old;
2. Patients treated and discharged from one of the four study sites with acute asthma (not simply for a prescription refill) during the study period;
3. Patients must have had a previous physician-diagnosis of asthma and an exacerbation diagnosed by the ED physician (e.g., past asthma history, recorded response to β-agonists in the ED, and increased asthma symptoms). In the event of a new diagnosis, the patient is still eligible for the study if the treating physician feels that the history is compatible with a diagnosis of asthma;
4. Patients must have evidence of airflow obstruction on presentation at the ED, defined as an FEV1 or PEF <80% of predicted;
5. Patients must not have a history of more than 20 pack-years of smoking;
6. All patients should have a PCP (FP, nurse practitioner or internist) with whom to follow-up or attempts will be made to find one for them.

Exclusion criteria:

These criteria ensure the exclusion of suspected COPD patients and patients who require different treatments:

1. Patients with asthma who are primarily cared for by a Respirologist/Pulmonologist;
2. Patients not seen by an emergency physician in the ED (e.g., direct referrals);
3. Physician diagnosis of acute COPD (e.g., failure of FEV1 or PEF to respond to ED treatment and a FEV1/FVC ratio ≤ 70%);
4. Radiologically confirmed pneumonia during the 10 days preceding trial entry;
5. Patients with an active history of bronchiectasis, cystic fibrosis, or lung cancer;
6. Clinically confirmed congestive heart failure at ED presentation;
7. Patients not able/unwilling to perform spirometry assessment;
8. Inability to provide informed consent or comply with the study protocol due to cognitive impairment, language barrier, or no contact details;
9. Patient has previously participated in the study;
10. Patients who in the opinion of the investigator are unsuitable for enrolment.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 367 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Relapses within 90 days after discharge | 90 days
  Any unscheduled medical visit to a walk-in clinic, family doctor's office or an emergency department resulting from the patient's perceived need for further asthma treatment within 90 days after discharge.

SECONDARY OUTCOMES:
Time to relapse | 90 days
  Time from Emergency Department (ED) discharge to first asthma relapse.
Primary care provider follow-up | 30 days
  A patient having a face-to-face meeting with their PCP within 30 days after discharge. Telephone interactions with the office will be classified as "no PCP follow-up".
Health related quality of life (HRQoL) | Baseline, 30 and 90 days
  A disease specific, validated instrument for asthma patients (AQLQ) will be used. We will also employ the EQ-5D.

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Rowe, MD, MSc, Principal Investigator — University of Alberta; Cristina Villa-Roel, MD, MSc, Principal Investigator — University of Alberta; Eddy Lang, MD, Principal Investigator — University of Calgary; Mohit Bhutani, MD, Principal Investigator — University of Alberta; Bjug Borgundvaag, MD, Principal Investigator — University of Toronto; Richard Leigh, MD, Principal Investigator — University of Calgary; Sumit Majumdar, MD, MSc, Principal Investigator — University of Alberta; Christopher McCabe, PhD, Principal Investigator — University of Alberta; Rhonda Rosychuk, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No